CLINICAL TRIAL: NCT01597232
Title: Effect of West China Perioperative Transfusion Score (WCPTS) on Red Blood Cells Transfusion in Patients Undergoing Major Surgery: a Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Clinic Trial for West China Perioperative Transfusion Score (WCPTS)
Acronym: WCPTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ren Liao, Associate Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WCPTS120508
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Transfusion Related Complications
Keywords: Transfusion trigger; Hemoglobin level

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Transfusion trigger based on WCPTS (Experimental): Determination of whether a patient need red blood cells transfusion or which hemoglobin level should be maintained is based on WCPTS.
  Interventions: Other: Transfusion trigger based on WCPTS
- Hemoglobin level 10g/dL (Active Comparator): The patient's hemoglobin level is maintained more than 10g/dL perioperatively.
  Interventions: Other: Maintenance of hemoglobin level more than 10g/dL
- Transfusion trigger based on experience (Active Comparator): Determination of whether a patient need red blood cell transfusion or which hemoglobin level should be maintained is base on the physician's experience.
  Interventions: Other: Transfusion trigger based on experience

INTERVENTIONS:
Other: Transfusion trigger based on WCPTS — Determination of whether a patient needs red blood cell transfusion or which hemoglobin level should be maintained is based on WCPTS
  Arms: Transfusion trigger based on WCPTS
Other: Maintenance of hemoglobin level more than 10g/dL — The patient's hemoglobin level is maintained more than 10g/dL perioperatively
  Arms: Hemoglobin level 10g/dL
Other: Transfusion trigger based on experience — Determination of whether the patient need red blood cell transfusion or which hemoglobin level should be maintained is based on the physician's experience
  Arms: Transfusion trigger based on experience

SUMMARY:
Guidelines for blood transfusion have been issued for years. According to these guidelines, red blood cells (RBCs) transfusion should be given when the hemoglobin level is less than 6g/dL or 7g/dL and is unnecessary when the level is more than 10g/dL. However, in all the guidelines, the determination of whether RBCs should be administered when the hemoglobin level is in the range of 6~10g/dL is based on the judgment from anesthesiologists or surgeons. Index of transfusion trigger for patients with hemoglobin level between 6g/dL and 10g/dL is necessary and important in clinical practice.

Based on the aim of blood transfusion that maintain the balance of oxygen supply and oxygen consumption, the investigators hypothesize that index of transfusion trigger for patients with hemoglobin level between 6g/dL and 10g/dL could be calculated by parameters including infusion rate of adrenalin for maintaining normal cardiac output, fraction of inspired oxygen, core temperature, and angina. To verify this hypothesis, the investigators present West China Perioperative Transfusion Score (WCPTS) for the trigger of transfusion according to the patient's history and monitoring parameters, and the investigators design a randomized controlled clinical trial to test this score.

DETAILED DESCRIPTION:
Surgery and trauma are the most common reasons for major blood loss, and blood transfusion provide guarantee for massive hemorrhagic surgery, especially orthopedic, cardiac, liver, and gynecologic procedures. On the other hand, blood transfusion is associated with many risks including hemolytic and nonhemolytic reactions, transfusion related acute lung injury (TRALI), and others. Besides, blood is insufficient worldwide. How to eliminate allogeneic blood transfusion is an important part in clinical practice.

Guidelines for blood transfusion have been issued for years. According to these guidelines, red blood cells (RBCs) transfusion should be given when the hemoglobin level is less than 6g/dL or 7g/dL and is unnecessary when the level is more than 10g/dL. However, in all the guidelines, the determination of whether RBCs should be administered when the hemoglobin level is in the range of 6~10g/dL is based on the judgment from anesthesiologists or surgeons. Index of transfusion trigger for patients with hemoglobin level between 6g/dL and 10g/dL is necessary and important in clinical practice.

Based on the aim of blood transfusion that maintain the balance of oxygen supply and oxygen consumption, the investigators hypothesize that index of transfusion trigger for patients with hemoglobin level between 6g/dL and 10g/dL could be calculated by parameters including infusion rate of adrenalin for maintaining normal cardiac output, fraction of inspired oxygen for maintaining spO2≧95%, core temperature, and angina.

Peri-Operative Transfusion Trigger Score, POTTS The initial score is 6. If a patient's cardiac output is normal without infusion of adrenalin, his spO2 could be maintained more than 95% with FiO2≤35%, his core temperature is less than 38℃, and he has no angina, his score is 6.

If a patient has one or more problems, including his normal cardiac output should be maintained by infusion of adrenalin with its rate ≤0.05μg/kg.min, or his spO2 is maintained more than 95% with 36~50% FiO2, or his core temperature is between 38℃ to 40℃, or chest pain due to exercise,manual labor,or excitement, his score should be added 1 point for each problem.

If a patient has one or more problems, including his normal cardiac output should be maintained by infusion of adrenalin with its rate >0.06μg/kg.min, or his spO2 is maintained more than 95% with >51% FiO2, or his core temperature is >40℃, or sudden onset of chest pain at rest, his score should be added 2 point for each problem.

The initial POTTS score is 6, and the patient's score is calculated by the sum of each item.

Score 6：The transfusion trigger is 6g/dL, and the the patient's Hemoglobin level should be maintained not less than 6g/dL.

Score 7：The transfusion trigger is 7g/dL, and the the patient's Hemoglobin level should be maintained not less than 7g/dL.

Score 8：The transfusion trigger is 8g/dL, and the the patient's Hemoglobin level should be maintained not less than 8g/dL.

Score 9：The transfusion trigger is 9g/dL, and the the patient's Hemoglobin level should be maintained not less than 9g/dL.

Score 10 or >10：The transfusion trigger is 10g/dL, and the the patient's Hemoglobin level should be maintained not less than 10g/dL.

For example, if a patient need ≤0.05μg/kg.min adrenalin to maintain his normal cardiac output (+1), his spO2 could be maintained more than 95% with FiO2≤35%, his core temperature is less than 38℃, and he has sudden onset of chest pain at rest (+2), his POTTS score could be calculated as 6 +1 (≤0.05μg/kg.min adrenalin to maintain his normal cardiac output) +2 (sudden onset of chest pain at rest), and his POTTS score is 9. That means this patient's transfusion trigger is 9g/dL, and his hemoglobin level should be maintained above 9 at this situation.

ELIGIBILITY:
Inclusion Criteria:

* Height of usual place of residence less than 2,500 metres above sea level
* Perioperative hemoglobin level possibly less than 10g/dL

Exclusion Criteria:

* Emergency operation
* ASA classification V or VI
* Serious blood system diseases
* Dysfunction of hemoglobin
* Hypervolemic hemodilution
* Tumor metastasis
* Psychopathy
* Refuse to sign consent

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1351 (Actual)
Dates: Start 2012-05-07 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Proportion of patients received red-cell | Up to 30 days postoperatively
  Proportion of patients received red-cell during peri-operative period
Composite of in-hospital complications and all-cause mortality by day-30 | Up to 30 days postoperatively
  Composite of in-hospital complications and all-cause mortality by day-30, and complications were defined as the serious ones that cause prolonged hospitalization, or life threatening, but could get recovery after intense treatment during hospitalization, or life threatening, resulting in significantly decreased quality of life.

SECONDARY OUTCOMES:
Incidences of in-hospital infectious complications. | Up to 30 days postoperatively
  Infectious complications were defined as infection at any site, such as pulmonary infection, urinary infection, etc.
Intensive Care Unit (ICU) admission rate | Up to 30 days postoperatively
  Proportion of patients with ICU admission
Length of hospital stay (LOS) | Up to 30 days postoperatively
  LOS was defined as the time frame from the day of hospital admission to discharge from the hospital (unit: days).
Hemoglobin level at different time points | Up to 30 days postoperatively
  Hb level was measured at the time points as follows: before operation, completion of operation, 24hrs after operation, before discharge, and before all red cells transfusion
Cost of transfusion and hospitalization | Up to 30 days postoperatively
  Allogeneic blood cost and total in-hospital cost
SF-8 questionnaire | Up to one year postoperatively
  Follow-up of quality of life during one year after operation
Healing status of surgical incision | Up to 30 days postoperatively
  Healing status of surgical incision was divided into grade Ⅰ, Ⅱ, and Ⅲ. Grade Ⅰ was defined as the wound healing nicely without any adverse reaction, grade Ⅱ was defined as the inflammatory wound without the need of re-incision, and grade Ⅲ was defined as the wound suppurated with the need of re-incision for clearance.
All-cause mortality during 1-year after operation | Up to one year postoperatively
  All-cause mortality by day-60, day-180 and 1-year after operation

CONTACTS AND LOCATIONS:
Overall Officials: Ren Liao, M.D., Study Director — Department of Anesthesiology, West China Hospital, Sichuan University; Jin Liu, M.D., Principal Investigator — Department of Anesthesiology, West China Hospital, Sichuan University
Locations (1):
- Department of Anesthesiology, West China Hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Liao R, Liu J, Zhang W, Zheng H, Zhu Z, Sun H, Yu Z, Jia H, Sun Y, Qin L, Yu W, Luo Z, Chen Y, Zhang K, Ma L, Yang H, Wu H, Liu L, Yuan F, Xu H, Zhang J, Zhang L, Liu D, Huang H. Individualized red-cell transfusion strategy for non-cardiac surgery in adults: a randomized controlled trial. Chin Med J (Engl). 2023 Dec 5;136(23):2857-2866. doi: 10.1097/CM9.0000000000002584. PMID 37052133